CLINICAL TRIAL: NCT04894019
Title: The Effect of Continuous Invasive Arterial Blood Pressure Monitoring on Postinduction Hypotension in Patients Having Major Surgery (AWAKE Trial): a Randomized Trial
Brief Title: Effect of Continuous Invasive Blood Pressure Monitoring on Postinduction Hypotension in Patients Having Major Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-10057-BO-ff
Record Dates: First submitted 2021-05-03; First posted 2021-05-20 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Blood Pressure; Perioperative Hypotension; Postinduction Hypotension

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous monitoring group (Experimental): In patients randomized to the continuous monitoring group, continuous invasive arterial blood pressure monitoring will be displayed on the patient monitor. The treating anesthesiologist will be blinded to intermittent blood pressure monitoring using upper-arm cuff oscillometry.
  Interventions: Device: Continuous invasive blood pressure monitoring
- Intermittent monitoring group (Active Comparator): In patients randomized to the intermittent monitoring group, intermittent blood pressure monitoring will be displayed on the patient monitor. The treating anesthesiologist is blinded to continuous invasive arterial blood pressure monitoring.
  Interventions: Device: Intermittent non-invasive blood pressure monitoring

INTERVENTIONS:
Device: Continuous invasive blood pressure monitoring — Continuous invasive blood pressure monitoring using an arterial catheter
  Arms: Continuous monitoring group
Device: Intermittent non-invasive blood pressure monitoring — Intermittent non-invasive blood pressure monitoring using upper-arm cuff oscillometry
  Arms: Intermittent monitoring group

SUMMARY:
This is a randomized trial (1) investigating whether continuous invasive arterial blood pressure monitoring using an arterial catheter reduces the area under a mean arterial pressure (MAP) of 65 mmHg within the first 15 minutes of anesthetic induction compared to intermittent arterial blood pressure monitoring using oscillometry in patients having major surgery under general anesthesia; and (2) investigating the effect of continuous invasive arterial blood pressure monitoring using an arterial catheter on cardiac output, stroke volume, and heart rate within the first 15 minutes of anesthetic induction compared to intermittent blood pressure monitoring using upper-arm cuff oscillometry in patients having major surgery under general anesthesia.

DETAILED DESCRIPTION:
not provided

ELIGIBILITY:
Inclusion Criteria:

Patients...

* at least 18 years of age
* scheduled for elective major surgery under general anesthesia that requires continuous invasive arterial blood pressure monitoring using a radial arterial catheter for clinical indications not related to the study

Exclusion Criteria:

* Clinical indication to insert the arterial catheter before anesthetic induction ("awake arterial catheter"; this is usually the case in patients with severe cardiovascular diseases, such as heart failure or left ventricular assist device)
* emergency surgery
* American Society of Anesthesiologists physical status classification V or VI
* need for femoral artery catheterization
* heart rhythms other than sinus rhythm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2021-05-16 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Area under a MAP of 65 mmHg within the first 15 minutes of anesthetic induction between the intervention and the control group. | during the induction period

SECONDARY OUTCOMES:
Effect of continuous invasive arterial blood pressure monitoring on cardiac output within the first 15 minutes of anesthetic induction between the intervention and the control group. | during the induction period
Effect of continuous invasive arterial blood pressure monitoring on stroke volume within the first 15 minutes of anesthetic induction between the intervention and the control group. | during the induction period
Effect of continuous invasive arterial blood pressure monitoring on heart rate within the first 15 minutes of anesthetic induction between the intervention and the control group. | during the induction period

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kouz K, Wegge M, Flick M, Bergholz A, Moll-Khosrawi P, Nitzschke R, Trepte CJC, Krause L, Sessler DI, Zollner C, Saugel B. Continuous intra-arterial versus intermittent oscillometric arterial pressure monitoring and hypotension during induction of anaesthesia: the AWAKE randomised trial. Br J Anaesth. 2022 Oct;129(4):478-486. doi: 10.1016/j.bja.2022.06.027. Epub 2022 Aug 23. PMID 36008202